CLINICAL TRIAL: NCT01592968
Title: A Prospective Phase III Randomized Trial to Compare Stereotactic Radiosurgery vs. Whole Brain Radiation Therapy for >/= 4 Newly Diagnosed Non-Melanoma Brain Metastases
Brief Title: Stereotactic Radiosurgery or Whole Brain Radiation Therapy in Treating Patients With Newly Diagnosed Non-melanoma Brain Metastases
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0884; NCI-2014-02058 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-2012-00850; 2011-0884 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Metastatic Malignant Neoplasm; Metastatic Malignant Neoplasm in the Brain
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Mental Status and Dementia Tests; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (SRS) (Experimental): Patients undergo SRS on day 1.
  Interventions: Other: Cognitive Assessment; Other: Quality-of-Life Assessment; Radiation: Stereotactic Radiosurgery
- Arm II (WBRT) (Experimental): Patients undergo WBRT 5 days per week (7 days per week for inpatients) for 2 weeks.
  Interventions: Other: Cognitive Assessment; Other: Quality-of-Life Assessment; Radiation: Whole-Brain Radiotherapy

INTERVENTIONS:
Other: Cognitive Assessment — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; stereotactic radiation therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
  Arms: Arm I (SRS)
Radiation: Whole-Brain Radiotherapy — Undergo WBRT
  Other Names: WBRT; whole-brain radiation therapy
  Arms: Arm II (WBRT)

SUMMARY:
This randomized phase III clinical trial compares stereotactic radiosurgery with whole brain radiation therapy to see how well they work in treating patients with non-melanoma cancer that has recently spread from the first location to the brain. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Stereotactic radiosurgery is a specialized type of radiation therapy that delivers a single, high dose of radiation directly to the tumor and may kill more tumor cells and cause less damage to normal tissue. Whole brain radiation therapy delivers a lower dose of radiation to the entire brain over several treatments. It is not yet known whether stereotactic radiosurgery works better than whole brain radiation therapy in treating patients with non-melanoma brain metastases. Stereotactic radiosurgery may also cause fewer thinking and memory problems than whole brain radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare local tumor control 4 months after treatment of patients with 4 to 15 intracranial non-melanoma metastases at the time of enrollment (=< 15 at time of treatment) treated with stereotactic radiosurgery (SRS) versus (vs.) whole brain radiation therapy (WBRT) in a prospective randomized trial.

II. To compare cognitive decline at 4 months defined as a significant decline (5 point decrease from baseline based on the reliable change index) in Hopkins Verbal Learning Test - Revised (HVLT-R) Total Recall after initial treatment with stereotactic radiosurgery (SRS) versus whole brain radiation therapy (WBRT) in patients with 4 to 15 non-melanoma brain metastases at the time of enrollment (=< 15 at time of treatment).

SECONDARY OBJECTIVES:

I. To determine local control and distant tumor control in the brain at 1, 4, 6, 9, and 12 months post treatment.

II. To determine overall survival in each treatment arm. III. To assess the pattern of neurocognitive change in memory at 1, 4, 6, 9, and 12 months post-treatment as well as executive function, attention, processing speed, and upper extremity fine motor dexterity.

IV. To evaluate the composite neurocognitive function score for both treatment arms.

V. To assess the pre-treatment factors of age, Karnofsky performance status (KPS), and extra-cranial disease in the predictive determination of local and distant control and neurocognitive outcome in each treatment arm.

VI. To assess the correlation between number of lesions and total volume of intracranial disease and neurocognitive outcome in each treatment arm.

VII. To compare time to initiation of systemic therapy from completion of radiotherapy between the two treatment arms.

VIII. To compare number of cycles of systemic therapy delivered following completion of radiation treatment in the two treatment arms.

IX. To document and descriptively compare post-treatment adverse side effects between the two treatment arms.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo SRS on day 1.

ARM II: Patients undergo WBRT 5 days per week (7 days per week for inpatients) for 2 weeks.

After completion of study treatment, patients are followed up at 1, 4, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have histological proof of malignant cancer, which is metastatic. Histological proof may be obtained from the primary tumor or another metastatic site. However, cytology alone is not an acceptable method of diagnosis.
* All patients must have greater than 3 but less than or equal to 15 metastatic lesions seen on a contrast enhancing MRI scan obtained not less than one month prior to study enrollment. Patients who are found to have up to 20 metastatic lesions at the time of treatment planning (on volumetric MRI once the head frame is in place) may still participate in the trial.
* All patients must be >/= 18 years of age.
* All patients must sign informed consent verifying that they are aware of the investigational nature of this study in keeping with the rules and policies of M.D. Anderson Cancer Center. The only acceptable consent form is the one attached at the end of this protocol, and it must have been approved and amended by the M.D. Anderson IRB.
* All patients must be eligible to have all lesions treated with SRS (i.e. maximum diameter of largest lesion < 3.5cm) as determined by the radiation oncologist .
* All patients must have adequate liver, renal, and hematologic function as defined by Aspartate Amino Transferase (AST)/Alanine Amino Transferase (ALT)/Alkaline Phosphatase < 2.5 times normal, calculated creatinine clearance > 30ml/min, and platelet count > 50,000.
* All patients should have normal coagulation, with international normalized ratio (INR) < 1.3 and able to withhold anti-coagulation medications a minimum of 24 hours prior to radiosurgery (or until INR normalizes), on the day of treatment and 24 hours after radiosurgery has concluded. Those patients getting WBRT may continue these medications.
* Patients can be undergoing concurrent systemic therapy, such as temozolomide, at the discretion of their treating oncologist.

Exclusion Criteria:

* Patients are excluded from this trial if they have melanoma, small cell carcinoma, lymphoma/leukemia, or germ cell histology (note, melanoma patients will be eligible for the sister trial to this trial which will be open simultaneously).
* Patients will be excluded if they have had prior surgical resection of metastatic cancer from the brain.
* Patients will be excluded if there is radiographic or CSF cytological evidence of leptomenengial disease.
* Patients will be excluded if they have had prior Whole Brain Radiotherapy (WBRT) or prophylactic cranial irradiation (PCI). Prior SRS or Gamma Knife radiosurgery to 1-3 metastases with minimum of (6) weeks to the most recent scan are allowed on protocol.
* Female patients of childbearing age will be excluded if they are pregnant as assessed by serum b-HCG or urine pregnancy test. A serum b-HCG test or urine pregnancy test will be performed no greater than 14 days prior to study registration.
* Patients will be excluded if they are unable to obtain an MRI scan.
* Patients will be excluded if they have < 4 lesions, or > 15 lesions at enrollment or > 20 lesions at the time of treatment (note: patients who qualify for enrollment based on having 4-15 lesions, but who are discovered to have up to 20 lesions on the volumetric MRI used for treatment planning will be allowed to continue on study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-08-02 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Local control rate | At 4 months
  Estimated for each treatment arm with 95% confidence intervals based on the estimates of time to local failure.
Proportion of patients with neurocognitive decline | At 4 months
  Defined as a decline of 5 or more points from baseline in Hopkins Verbal Learning Test - Revised (HVLT-R) score. Estimated for each treatment arm with 95% confidence intervals based on the estimates of time to neurocognitive decline.

SECONDARY OUTCOMES:
Time to local failure | Up to 12 months
  Estimated using the product-limit estimator for each treatment arm. The logrank test stratified by the stratification factors will be used at randomization to compare the 2 treatment arms with respect to the time to local failure.
Cumulative incidence of local failure | Up to 12 months
  Estimated with death as a competing event.
Time to neurocognitive decline | Up to 12 months
  Measured by Hopkins Verbal Learning Test - Revised (HVLT-R) score. Estimated for each treatment arm using the product limit estimator of Kaplan and Meier. The logrank test stratified by the stratification factors will be used at randomization to compare the 2 treatment arms with respect to the time to neurocognitive decline.
Cumulative incidence of neurocognitive decline | Up to 12 months
  Estimated with death as a competing event.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org